CLINICAL TRIAL: NCT01254526
Title: A Phase Ib, Open-Label, Dose-Escalation Study of the Safety and Pharmacology of GDC-0980 in Combination With Paclitaxel With or Without Bevacizumab in Patients With Locally Recurrent or Metastatic Breast Cancer
Brief Title: Study of the Safety and Pharmacology of GDC-0980 in Combination With Paclitaxel With or Without Bevacizumab in Patients With Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIM4880g; GO00882 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-12-01; First posted 2010-12-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 1-(4-((2-(2-aminopyrimidin-5-yl)-7-methyl-4-morpholinothieno(3,2-d)pyrimidin-6-yl)methyl)piperazin-1-yl)-2-hydroxypropan-1-one; Bevacizumab; Paclitaxel

ARMS (2):
- A (Experimental)
  Interventions: Drug: GDC-0980; Drug: paclitaxel
- B (Experimental)
  Interventions: Drug: GDC-0980; Drug: bevacizumab; Drug: paclitaxel

INTERVENTIONS:
Drug: GDC-0980 — Oral repeating dose
Drug: bevacizumab — Intravenous repeating dose
  Arms: B
Drug: paclitaxel — Intravenous repeating dose

SUMMARY:
This is an open-label, multicenter, Phase Ib dose-escalation study to assess the safety, tolerability, and pharmacokinetics of GDC-0980 administered with taxane-based chemotherapy regimens utilized in patients with locally recurrent or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Locally recurrent or metastatic breast cancer, not amenable to resection with curative intent
* For Arm C: Overexpression of HER2
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Adequate hematologic and organ function
* Evaluable or measurable disease per RECIST (Response Evaluable Criteria in Solid Tumors)
* Female patients of childbearing potential must use an acceptable method of contraception to prevent pregnancy and to continue its use for the duration of the study

Exclusion Criteria:

* Prior anti-cancer therapy of more than two regimens of systemic cytotoxic chemotherapy for advanced or metastatic breast cancer
* Prior anti-cancer therapy (e.g., chemotherapy, biologic therapy, or hormonal therapy) within a specified timeframe of the first dose of study treatment
* History of Type 1 or Type 2 diabetes requiring regular medication
* History of clinically significant cardiac or pulmonary dysfunction
* History of malabsorption syndrome or other condition that would interfere with enteral absorption
* Any condition requiring full-dose anticoagulants
* Leptomeningeal disease as a manifestation of cancer
* Active infection requiring IV antibiotics
* Active autoimmune disease that is not controlled by non-steroidal anti-inflammatory drugs, inhaled steroids, or the equivalent of <= 10 mg/day of prednisone
* Known clinically significant history of liver disease, including active viral, alcoholic, or other hepatitis, or cirrhosis
* Known HIV infection
* Known untreated or active CNS metastases
* Pregnancy, lactation, or breastfeeding
* Major surgical procedure, open biopsy, or significant traumatic injury within a within a specified timeframe of the first dose of study treatment

For Arm B:

* Uncontrolled hypertension, complication from hypertension, myocardial infarctions, unstable angina, vascular disease or stroke within a specified timeframe of the first dose of study treatment
* Evidence of bleeding diathesis or significant coagulopathy including hemoptysis within a specified timeframe of the first dose of study treatment
* History of abdominal conditions (e.g., fistula, perforation, obstruction) that would preclude use of bevacizumab
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities (DLTs) | Through Day 22
Incidence, nature, and severity of adverse events | Through study completion, up to 1 year, or early discontinuation

SECONDARY OUTCOMES:
Pharmacokinetic parameters of GDC-0980, paclitaxel and bevacizumab (including total exposure, maximum and minimum plasma concentration, time to maximum observed plasma concentration, plasma half-life) | Through Day 22
Duration of response | Assessed at periodic intervals until study completion, up to 1 year, or early discontinuation
Progression-free survival (PFS) | Assessed at periodic intervals until study completion, up to 1 year, or early discontinuation
Objective tumor response | Assessed at periodic intervals until study completion, up to 1 year, or early discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Lauchle, M.D., Study Director — Genentech, Inc.
Locations (3):
- United States (2):
  - Boston, Massachusetts
  - Nashville, Tennessee
- Leuven, Belgium